CLINICAL TRIAL: NCT03060265
Title: Protective Analgesia in Caesarean Section Using Intravenous Paracetamol: A Prospective Randomised Controlled Trial
Brief Title: Protective Analgesia in Caesarean Section Using Intravenous Paracetamol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, Director of Anesthesia Department, Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: BnaiZionMC-16-MS-003
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Analgesia
Keywords: multimodal analgesia; paracetamol; cesarean section
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Active Comparator): Paracetamol Braun Germany 1 gram in 100ml normal saline, one dose IV
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): 100ml normal saline, one dose IV
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Paracetamol — Administrating Paracetamol IV pre-cesarean section
  Other Names: Acamol
  Arms: Paracetamol
Drug: PLACEBO — Administrating SALINE IV pre-cesarean section
  Other Names: SALINE
  Arms: Placebo

SUMMARY:
Protective analgesia in caesarean section using intravenous paracetamol: A prospective randomised controlled trial. Cesarean section a common surgical procedure in women. The parturients undergoing CS experience severe to moderate postoperative pain. Pain relief is very important to the patient as it causes discomfort which affects hemodynamic intraoperative and increases the risk of postoperative complications. Analgesia is crucial to postoperative recovery.

Aims: To investigate the efficacy of combined administration of paracetamol, as protective multimodal analgesia, and standard spinal anesthesia in the reduction of postoperative pain following cesarean section.

Sixty adult Parturients undergoing CS will participate in a single-centered, randomized, double-blinded, placebo-controlled trial divided into 2 groups 30 each. The intervention group will receive 1 gr of intravenous paracetamol in 100 ml normal saline only 15 minutes prior to spinal anesthesia induction. The control group will receive 100 ml normal saline IV identical in size and shape and manner to the experimental group, 15 minutes prior to induction of spinal anesthesia. We will measure postoperative Visual Analog Scale (VAS) pain score, postoperative time to analgesia in PACU and number of postoperative analgesic doses within 24 hours.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of most common surgical procedure in women. Parturients undergoing CS, experience severe to moderate postoperative pain. Pain after CS may impair the ability of mother to care and feed her child, early ambulation, and discharge. About 12.3% of parturients experience pain scores enough to affect infant care up to 6 months after CS.

All of perioperative stress effects, before delivery of the baby, such as, skin incision, need various approaches of treatment, which may include systemic and neuraxial analgesia.

Surgical trauma causes immediate changes in both peripheral and central nervous systems, leading to augmentation of pain perception in the final destination - the cerebral cortex. The surgical incision induces secretion of cyclooxygenase-2 (COX-2), which increases the production of prostaglandins (PGs), and which in turn excites peripheral nociceptors. These special pain fibers not only transmit the pain signal to the central nervous system, but also amplify tissue sensitivity to the surgical trauma, giving rise to the phenomenon known as "local hyperalgesia".

Improper pain control during the perioperative period leads to complications, which may affect the outcome of CS. Pain relief is very important to the patient as the pain causes discomfort which affects hemodynamic intraoperative and increases the risk of postoperative complications as atelectasis, ineffective, coughing and inadequate ventilation. Adequate pain control is essential not only intraoperatively, but also in immediate postoperative period to cover long time period postoperatively. The major role of intra- or post-operative management of pain is to reduce the dose of medication and to lessen side-effects, while providing adequate analgesia. This role may best be accomplished with multimodal protective analgesia or preemptive analgesia. Protective multimodal analgesia term is described as any intraoperative analgesic agents able to control pain-induced sensitization of the central nervous system. Preemptive analgesia had been defined as an antinociceptive treatment, starts before surgery that to prevent establishment of altered central afferent input from injuries and its goal is to decrease pain by timing the analgesic's peak pharmacodynamic effect with anticipated onset of pain or peak pain response.

Protective analgesia is distinguished from pre-emptive analgesia in that it focuses less on the treatment and on the relatively timing and the anesthetic intervention but rather more on the mechanisms of action. Protective analgesia aims to decrease the impact of the nociceptive barrage associated with noxious pre-operative, intra-operative, and/or post-operative events/stimuli.

Systemic opioids either intra- or post-operatively have potential of serious adverse reactions or risks for neonate and they act on opioid center in central nervous system. Paracetamol (Acetaminophen) is mostly used for treating pain and fever, typically for mild to moderate pain. In combination with opioid agents, paracetamol is used for more severe pain such as in cases of cancer and after surgery.

Paracetamol is devoid of risks related to opioid and acts at both central and peripheral points of the pain pathway, by direct inhibition of N-methyl-D-Aspartate receptors and inhibition of the cyclooxygenase 2 (COX-2) pathway.

Spinal anesthesia using local anesthetics combined with opioids affects the transmission, modulation and modification stages of nociceptive afferent impulses and its analgesic qualities are superior to local anesthesia alone.

Study where paracetamol as pre-emptive analgesia was compared to placebo in paediatric after tonsillectomy patients, found that pain score was lower in the experimental group.

In patients undergoing lower extremity surgery with spinal anesthesia, protective acetaminophen may enhance analgesia and decrease postoperative analgesic consumption.

To our knowledge, no studies have investigated the combined use of paracetamol with spinal anesthesia/analgesia for pre, intra and postoperative multimodal pain protection in parturients undergoing cesarean section.

The aim of our study is therefore; to assess the efficacy of combined administration of paracetamol and standard spinal anesthesia in the reduction of postoperative pain following cesarean section.

Materials and Methods

Study population

A single-center, prospective, randomized, double-blind, placebo-controlled study will be conducted at Bnai-Zion Medical Center, Haifa, Israel (following the approval and according to the regulations of the Helsinki Committee).

Inclusion criteria consist of parturient age between 18 and 40 years, a maximal American Society of Anesthesiologists (ASA) Score of II, parturients undergoing first elective cesarean section.

Exclusion criteria consist of current or previous chronic NSAID or opioid treatment, liver or renal insufficiency, asthma, cardiovascular disease, allergy to paracetamol or other NSAIDs. Parturients with ASA III, IV and whom past a spinal anesthesia failure will be also excluded from the study. All parturient participants will provide written informed consent.

Study protocol

Parturients will be blindly and randomly allocated to 2 groups, consisting of 30 patients each, randomization will be performed with a computer-generated. The experimental group participants will be treated with 1 gr paracetamol (under the brand name Paracetamol® B. Braun, Germany) intravenous provided in 100 ml normal saline in a single intravenous dose in a double-blind mode. Where in the control placebo group participants will be provided with the same bag of 100 ml normal saline medication free. Each bag contains the patient allocation number, the package identification number, the bag type (A for paracetamol or B for placebo). Separate sealed envelopes will be provided to the investigator to be opened in the event of a serious adverse event. The treatment will be conducted in both groups at the same time, 15 minutes prior to spinal anesthesia induction. [The control group will receive 100 ml normal saline identical in size and shape to the treatment drug, 15 minutes prior to induction of spinal anesthesia.] All parturients will receive spinal anesthesia using 10-12mg of bupivacaine for local anesthesia and 25μg of fentanyl. The agents will be administered by senior anesthesiologists, who are not involved in data collection. The same surgical team will perform all cesarean sections.

Data collection

In addition to demographic data parturient age, weight, the following parameters will be collected:

* Heart rate, systolic blood pressure, diastolic blood pressure, and peripheral oxygen saturation.
* The pain intensity level presented in VAS scale (0- none, 10-the worst imaginable pain) will be estimated and marked at arrival in PACU ,2, 4, 8, 12 and 24 hours postoperatively will be estimated.
* Postoperative time to first administration of analgesic dose (Time-to-Analgesia; TTA) will be noted.
* Number of analgesic doses administered within the first 24 hours after surgery.
* When in the PACU and in surgical ward, the VAS score ≥4, 1-3 mg of morphine IV in titration boluses will be administrated.
* Pain relief will be evaluated and recorded on a five-point scale (0 - none, 1 - a little, 2 - some, 3- a lot, and 4- complete). Analgesic agents will be titrated till pain score reaches zero or stage 1 (a little pain).
* Side effects such as local pain, nausea, vomiting, hypotension, be recorded.

Power and statistical analysis

A sample size of 30 parturients by group is calculated to detect a significant difference of 20% or more in intraoperative opioid consumption with a power of 100% two-tailed and a significant level of 5% (alpha of 0.05) corresponding to level of confidence 95%. Data will be reported as mean ± SD and counts (numbers).

With the following assumptions:

* A 30% difference in postoperative analgesic doses
* A 40 minutes difference for TTA
* A 30 % difference in the postoperative VAS score. Statistical assessment includes analysis of Student's t-test for continuous data and VAS pain data. Fisher's exact t-test will be used to analyze nominal data. P < 0.05 will be considered to be significant for all tests. All analyses will be performed using the SPSS statistical software, version 15 (SPSS Inc.; Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Parturient age between 18 and 40 years,
* A maximal American Society of Anesthesiologists (ASA) Score of II,
* Parturients undergoing first elective cesarean section.

Exclusion Criteria:

* Current or previous chronic NSAID or opioid treatment, liver or renal insufficiency, asthma, cardiovascular disease, allergy to paracetamol or other NSAIDs.
* Parturients with ASA III, IV and whom spinal anesthesia failure will be also excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The pain intensity level | 24 hours
  measured by VAS score The pain intensity level presented in VAS scale (0- none, 10-the worst imaginable pain) will be estimated and marked at arrival in PACU ,2, 4, 8, 12 and 24 hours postoperatively will be estimated.

SECONDARY OUTCOMES:
side effects | 24 hours
  Side effects such as local pain, nausea, vomiting, hypo tension, be recorded.
Postoperative time to administration of first analgesic dose (Time-to-Analgesia; TTA). | 24 hours
  measuring time in mins or hours
Number of analgesic doses administered in the first 24 hours after surgery. | 24 hours
  recording the administration of analgesic doses in number

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, Prof, Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: No